CLINICAL TRIAL: NCT03549494
Title: Effect of Ocoxin®-Viusid® Nutritional Supplement on the Quality of Life of Patients With Advanced Stomach Cancer and Esophagogastric Junction. Phase II Clinical Trial.
Brief Title: Evaluation of Ocoxin®-Viusid® in Advanced Stomach Cancer and Gastric Esophagogastric Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-8
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stomach Neoplasm; Gastrointestinal Neoplasms; Digestive System Neoplasm; Esophageal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Disease; Digestive System Disease; Esophageal Diseases; Stomach Diseases; Esophagogastric Junction Disorder
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Gastrointestinal Diseases; Digestive System Diseases; Esophageal Diseases; Stomach Diseases | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocoxin-Viusid® (Experimental)
  Interventions: Dietary Supplement: Ocoxin-Viusid®

INTERVENTIONS:
Dietary Supplement: Ocoxin-Viusid® — Ocoxin-Viusid group (Experimental). Oral solution of Ocoxin-Viusid (vials of 30 ml), at a rate of 60 ml daily (1 vial every 12 hours), administrado preferably administered after breakfast and dinner. The product will dilute in water, milk or juice. The treatment will have a period of 19 weeks, starting 2 weeks before the onco-specific treatment with FOLFOX chemotherapy and will end 3 weeks after the end of the sixth cycle of chemotherapy. QT FOLFOX will be prescribed intravenously every 14 days for 6 cycles as follows: Oxaliplatin (85 mg x m2) on day 1 Folinic acid (200 mg x m2) on day 1 and 2 5 Fluoracil (400 mg x m2, bolus) on day 1 and 2 5 Fluoracil (600 mg x m2, continuous infusion) on day 1 and 2

SUMMARY:
Our main objective is to evaluate the effect of Ocoxin-Viusid on the quality of life of patients with advanced stomach cancer and esophagogastric junction. The Ocoxin-Viusid nutritional supplement is expected to improve quality of life and tolerance to treatment with Chemotherapy.

DETAILED DESCRIPTION:
* To evaluate the effect of Ocoxin-Viusid on the quality of life of patients
* To evaluate the toxicity of Ocoxin-Viusid in combination with chemotherapy (QT).
* To assess the influence of Ocoxin-Viusid on tolerance to treatment with chemotherapy.
* Identify the changes that occur in the nutritional status of patients receiving the supplement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cyto-histological diagnosis of stomach adenocarcinoma and gastric esophageal junction in stages III and IV, which are tributaries of the FOLFOX chemotherapy scheme.
2. Patients of any sex with age ≥ 18 years.
3. Patients with clinical status according to Karnofsky index ≥ 70%.
4. Patients with life expectancy ≥ 3 months.
5. Clinically fit patients to receive the FOLFOX chemotherapy scheme.
6. Patients who have signed informed consent for the investigation.
7. Patients with laboratory parameters within normal limits that do not contraindicate the administration of chemotherapy: hemoglobin ≥ 90 g / l, total leukocyte count ≥ 3.0 x 109 / L, absolute neutrophil count> 1.5 x 109 / L, platelet count> 100 x 109 / L, total bilirubin ≤ 1.5 times the upper limit of the normal range established in the institution, TGO / TGP ≤2.5 times the upper limit of the normal range established in the institution, creatinine within the limits normal of the institution.
8. Patients of childbearing age with negative pregnancy test and use appropriate contraceptive methods such as intrauterine devices, barrier or tubal ligation methods, hormonal contraceptives. In the case of male sex (vasectomy, use of condoms) while the treatment lasts.

Exclusion Criteria:

1. Patients with stomach cancer and gastric esophageal junction in stages III and IV, tributaries of surgical treatment and / or radiotherapy.
2. Patients who are being treated with another product under investigation.
3. Patients with known hypersensitivity to any component of the investigational product.
4. Patients with known hypersensitivity to any component of the Chemotherapy (FOLFOX).
5. Patients with acute allergic states or history of severe allergic reactions.
6. Patients with acute, chronic, or inflammatory decompensated infectious diseases.
7. Patients with brain metastases.
8. Patients with psychiatric disorders that make it difficult to collect information, treatment or follow-up.
9. Patients in the period of breast-feeding or puerperium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 5 months
  Karnofsky index (Score of 0-100 points at intervals of 10).
Quality of Life | 5 months
  EORTC QLQ-C30 (score of every item and global score)
Quality of Life | 5 months
  EORTC QLQ-STO22 if gastric cancer (score of every item and global score)
Quality of Life | 5 months
  EORTC QLQ-OG25 if is a gastric esophagus union cancer (score of every item and global score)

SECONDARY OUTCOMES:
Nutritional Status | 5 months
  Body mass Index calculated by Weight/(Height*Height), the weight expressed in Kg and, the height expressed in meters.
Chemotherapy Tolerance | 5 months
  Adverse Reactions (It will consider the compliance to the Chemotherapy treatment in terms of time and doses plan and, it will classify in "Yes, No").
Adverse Events-AE | 5 months
  AE will be measured as: - Type of AE (Description of the EA that is presented) - Causal Agent (QT, Oncoxin -Viusid, Other) - Seriousness of the AE (Serious, Not serious) - Intensity of the AE (Mild, Moderate, Severe, Life-threatening consequences, Death, according to the Common Criteria of Adverse Event Terminology (CTCAE) version 4.0) - Duration of the AE (Difference between the start and end date of the event) - Causal relationship (Very likely/Definitive, Probable, Possible, Unlikely, Not related, Not assessable/Not classifiable according to the WHO classification) - Attitude towards treatment (No change, Modification of doses, Temporary interruption, Definitive interruption)
Results of laboratory tests | 5 months
  Hematological (hemoglobin, platelets, total leukocytes, CAN) and Blood chemistry (AST, ALT, total bilirubin, creatinine, glycemia, albumin, total proteins, alkaline phosphatase) .The values will be recorded according to the units established for each test, reporting as normal, abnormal, not clinically significant, abnormal clinically significant and not performed, according to the normality ranges of the institution)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology and Radiobiology (INOR), Havana, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Lamson DW, Brignall MS. Antioxidants in cancer therapy; their actions and interactions with oncologic therapies. Altern Med Rev. 1999 Oct;4(5):304-29. PMID 10559547
- [Background] Lamson DW, Brignall MS. Natural agents in the prevention of cancer, part two: preclinical data and chemoprevention for common cancers. Altern Med Rev. 2001 Apr;6(2):167-87. PMID 11302780
- [Background] Block KI, Koch AC, Mead MN, Tothy PK, Newman RA, Gyllenhaal C. Impact of antioxidant supplementation on chemotherapeutic toxicity: a systematic review of the evidence from randomized controlled trials. Int J Cancer. 2008 Sep 15;123(6):1227-39. doi: 10.1002/ijc.23754. PMID 18623084
- [Background] Prasad KN, Hernandez C, Edwards-Prasad J, Nelson J, Borus T, Robinson WA. Modification of the effect of tamoxifen, cis-platin, DTIC, and interferon-alpha 2b on human melanoma cells in culture by a mixture of vitamins. Nutr Cancer. 1994;22(3):233-45. doi: 10.1080/01635589409514349. PMID 7877893
- [Background] Rodrigues MJ, Bouyon A, Alexandre J. [Role of antioxidant complements and supplements in oncology in addition to an equilibrate regimen: a systematic review]. Bull Cancer. 2009 Jun;96(6):677-84. doi: 10.1684/bdc.2009.0886. French. PMID 19493854
- [Background] Bardia A, Tleyjeh IM, Cerhan JR, Sood AK, Limburg PJ, Erwin PJ, Montori VM. Efficacy of antioxidant supplementation in reducing primary cancer incidence and mortality: systematic review and meta-analysis. Mayo Clin Proc. 2008 Jan;83(1):23-34. doi: 10.4065/83.1.23. PMID 18173999
- [Background] Hernandez-Unzueta I, Benedicto A, Olaso E, Sanz E, Viera C, Arteta B, Marquez J. Ocoxin oral solution(R) as a complement to irinotecan chemotherapy in the metastatic progression of colorectal cancer to the liver. Oncol Lett. 2017 Jun;13(6):4002-4012. doi: 10.3892/ol.2017.6016. Epub 2017 Apr 10. PMID 28599406
- [Background] Hernandez-Garcia S, Gonzalez V, Sanz E, Pandiella A. Effect of Oncoxin Oral Solution in HER2-Overexpressing Breast Cancer. Nutr Cancer. 2015;67(7):1159-69. doi: 10.1080/01635581.2015.1068819. Epub 2015 Aug 4. PMID 26241555
- [Background] Lagergren P, Fayers P, Conroy T, Stein HJ, Sezer O, Hardwick R, Hammerlid E, Bottomley A, Van Cutsem E, Blazeby JM; European Organisation for Research Treatment of Cancer Gastrointestinal and Quality of Life Groups. Clinical and psychometric validation of a questionnaire module, the EORTC QLQ-OG25, to assess health-related quality of life in patients with cancer of the oesophagus, the oesophago-gastric junction and the stomach. Eur J Cancer. 2007 Sep;43(14):2066-73. doi: 10.1016/j.ejca.2007.07.005. Epub 2007 Aug 15. PMID 17702567
- [Background] Gomez EV, Perez YM, Sanchez HV, Forment GR, Soler EA, Bertot LC, Garcia AY, del Rosario Abreu Vazquez M, Fabian LG. Antioxidant and immunomodulatory effects of Viusid in patients with chronic hepatitis C. World J Gastroenterol. 2010 Jun 7;16(21):2638-47. doi: 10.3748/wjg.v16.i21.2638. PMID 20518086